CLINICAL TRIAL: NCT04399928
Title: A Prospective, Multicenter, Non-randomized, Clinical Outcomes Study of the R3◊ Acetabular System in Patients With Degenerative Hip Disease
Brief Title: EU Safety and Efficacy Study Regarding the R3 Acetabular Hip System
Status: Completed | Type: Observational
Sponsor: Smith & Nephew Orthopaedics AG (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Other Study IDs: SR 16-4845-15 (R11019)
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2022-05

CONDITIONS: Degenerative Joint Disease
Keywords: Degenerative joint disease; Total Hip Arthroplasty
MeSH Terms: conditions — Joint Diseases | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Device: Total Hip Arthroplasty — Total hip arthroplasty with the R3 Acetabular Hip system.

SUMMARY:
The objective of this study is to determine the long-term safety and effectiveness from the R3 Acetabular Hip System. The study hypothesis is that implant survivorship of the R3 cup is at least 97% at 3 years, 95% at 5 years, 93% at 7 years, and 90% at 10 years follow-up.

DETAILED DESCRIPTION:
This is a multicenter prospective observational post-market clinical follow-up study that will include 500 patients who will have total hip replacement with the R3 Acetabular System and either cemented or cementless hip stem.

Effectiveness will be assessed by comparison of changes in parameters contained in the HOOS questionnaire and based upon incidence of revision and change in Harris Hip Score and UCLA Rating. Safety will be measured by assessing all adverse events experienced by patients from study enrolment through to study completion.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following characteristics for inclusion in the study.

* Patient is 18-75 years old and he/she is skeletally mature
* Patient requires primary total hip arthroplasty due to non-inflammatory degenerative joint disease (e.g. osteoarthritis, post-traumatic arthritis, avascular necrosis, dysplasia/DDH or inflammatory joint disease (e.g., rheumatoid arthritis)
* Patient has met an acceptable preoperative medical clearance and is free from or treated for cardiac, pulmonary, hematological, etc., conditions that would pose excessive operative risk
* The patient is willing to comply the follow-up schedule

Exclusion Criteria:

Subjects with any of the following characteristics must be excluded from the participation in the study.

* Patient has active infection or sepsis (treated or untreated)
* Patient is a prisoner or has an emotional or neurological condition that would pre-empt their ability or unwillingness to participate in the study including mental illness, mental retardation, linguistic insufficiencies (i.e. immigrants), or drug/alcohol abuse.
* Patients with acute hip trauma (femoral neck fracture)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This clinical study can fulfill its objectives only if appropriate subjects are enrolled. All relevant medical and non-medical conditions should be taken into consideration when deciding whether a particular patient is suitable. Subjects will be enrolled consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 479 (Actual)
Dates: Start 2009-05-18 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Remes, Associate Professor, Principal Investigator — University of Helsinki
Locations (8):
- AZ Nikolaas, Sint-Niklaas, Moerlandstraat 1, Belgium
- Hvidovre University Hospital, Hvidovre, Denmark
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - TYKS Turku University Hospital, Turku
- Knappschaftskrankenhaus Püttlingen, Püttlingen, Germany
- Medisch Centrum Alkmaar, Alkmaar, Netherlands
- University Hospital La Paz, Madrid, Spain
- The Royal Orthopaedic Hospital, NHS Foundation Trust, Birmingham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The data from one (1) enrolled hip (1 participant) were entirely removed due to questions regarding the validity of the participant's consent.
Units Other Than Participants: hips
Groups:
- R3™ Acetabular System: Total hip replacement with the R3™ Acetabular System (cemented or cementless hip stem)
Period: Overall Study
Arm/Group | R3™ Acetabular System
Started | 478; 501 hips
Completed | 350; 366 hips
Not Completed | 128; 135 hips

BASELINE CHARACTERISTICS:
Units Other Than Participants: hips
Arm/Group | R3™ Acetabular System
Number analyzed (Participants) | 478
Number analyzed (hips) | 501
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (9.02)
Sex: Female, Male [Count of Units; unit: hips]
  Female | 284
  Male | 217
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: hips]
  Netherlands | 38
  Belgium | 97
  Finland | 142
  Denmark | 104
  United Kingdom | 49
  Germany | 38
  Spain | 33
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.0 (5.11)

OUTCOME MEASURES:

1. Primary Outcome: Implant Survivorship
Description: Implant survivorship by 10 years post study procedure measured by Kaplan-Meier survival rate. Implant survival determined by no revision required for any reason. A revision is a surgical procedure of the study hip where one or more of the study components are removed and replaced with new implants.
Time Frame: up to 10 years post-operatively
Population: Safety Analysis Population (SAF) included participants enrolled and implanted with the study device with data collected for the time frame indicated.
Measure: Number (95% Confidence Interval); unit: percentage of hips
Units Other Than Participants: hips
Arm/Group | R3™ Acetabular System
Number analyzed (Participants) | 478
Number analyzed (hips) | 501
percentage of hips | 0.89 [0.865 to 0.923]

2. Secondary Outcome: Patient Reported Outcome (PRO): Hip Disability and Osteoarthritis Outcome Score (HOOS)
Description: HOOS is a measurement of function and outcomes of daily living that ranges from 0 to 100 where 0 indicated extreme symptoms (i.e., worse outcome) and 100 indicated no symptoms (i.e., better outcome).
Time Frame: Pre-operative, 3 months, 1 years, 3 years, 5 years, 7 years, 10 years
Population: Full Analysis Set (FAS) population included participants enrolled and implanted with the study device with data available from at least one post-operative assessment for the time frame indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: hips
Arm/Group | R3™ Acetabular System
Number analyzed (Participants) | 429
Number analyzed (hips) | 449
score on a scale
  Pre-operative | 37.8 (16.16)
  3 Months: number analyzed (Participants) | 419
  3 Months: number analyzed (hips) | 436
  3 Months | 83.2 (12.39)
  1 Year: number analyzed (Participants) | 395
  1 Year: number analyzed (hips) | 417
  1 Year | 88.1 (12.48)
  3 Years: number analyzed (Participants) | 376
  3 Years: number analyzed (hips) | 396
  3 Years | 87.9 (12.22)
  5 Years: number analyzed (Participants) | 319
  5 Years: number analyzed (hips) | 337
  5 Years | 88.0 (13.76)
  7 Years: number analyzed (Participants) | 299
  7 Years: number analyzed (hips) | 316
  7 Years | 87.5 (12.43)
  10 Years: number analyzed (Participants) | 305
  10 Years: number analyzed (hips) | 321
  10 Years | 89.3 (10.69)

3. Secondary Outcome: Patient Reported Outcome (PRO): Modified Harris Hip Score (mHHS)
Description: The mHHS scoring assessment ranges from 0 (worst) to 100 (best). Scores assessed during the pre-operative, 3-year, 5-year, 7-year and 10-year visit.
Time Frame: Pre-operative, 3 months, 1 years, 3 years, 5 years, 7 years, 10 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: hips
Arm/Group | R3™ Acetabular System
Number analyzed (Participants) | 454
Number analyzed (hips) | 475
score on a scale
  Pre-operative: number analyzed (Participants) | 452
  Pre-operative: number analyzed (hips) | 473
  Pre-operative | 51.5 (14.25)
  3 Months | 85.5 (13.78)
  1 Year: number analyzed (Participants) | 420
  1 Year: number analyzed (hips) | 442
  1 Year | 92.2 (11.67)
  3 Years: number analyzed (Participants) | 388
  3 Years: number analyzed (hips) | 408
  3 Years | 92.2 (10.91)
  5 Years: number analyzed (Participants) | 338
  5 Years: number analyzed (hips) | 357
  5 Years | 93.1 (10.93)
  7 Years: number analyzed (Participants) | 315
  7 Years: number analyzed (hips) | 333
  7 Years | 92.3 (10.90)
  10 Years: number analyzed (Participants) | 272
  10 Years: number analyzed (hips) | 285
  10 Years | 92.5 (10.71)

4. Secondary Outcome: Patient Reported Outcome (PRO): University of California, Los Angeles (UCLA) Rating
Description: UCLA Activity Score is a measure of physical activity levels in participants undergoing total joint arthroplasty. The scale ranges from 1 to 10 with higher scores indicating greater physical function (i.e., a better outcome).
Time Frame: Pre-operative, 3 months, 1 years, 3 years, 5 years, 7 years, 10 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: hips
Arm/Group | R3™ Acetabular System
Number analyzed (Participants) | 466
Number analyzed (hips) | 488
score on a scale
  Pre-operative | 3.4 (1.35)
  3 Months: number analyzed (Participants) | 464
  3 Months: number analyzed (hips) | 486
  3 Months | 5.2 (1.56)
  1 Year: number analyzed (Participants) | 422
  1 Year: number analyzed (hips) | 444
  1 Year | 6.1 (1.58)
  3 Years: number analyzed (Participants) | 398
  3 Years: number analyzed (hips) | 419
  3 Years | 6.1 (1.66)
  5 Years: number analyzed (Participants) | 342
  5 Years: number analyzed (hips) | 361
  5 Years | 6.1 (1.66)
  7 Years: number analyzed (Participants) | 318
  7 Years: number analyzed (hips) | 336
  7 Years | 5.7 (1.61)
  10 Years: number analyzed (Participants) | 314
  10 Years: number analyzed (hips) | 330
  10 Years | 5.6 (1.71)

5. Secondary Outcome: Radiographic Findings: Atrophy
Description: Number of participant hips with radiographic findings for atrophy indicated with a 'No', 'Yes', or 'N/A' (response not available) response at 1 year, 3 years, 5 years, 7 years, & 10 years for the following:
  * Atrophy in any Cup Zones
  * Atrophy in any Stem Zones
Time Frame: 1 years, 3 years, 5 years, 7 years, 10 years
Population: Participants enrolled and implanted with the study device with data collected from at least one post-operative assessment for the time frame indicated.
Measure: Count of Units; unit: hips
Units Other Than Participants: hips
Arm/Group | R3™ Acetabular System
Number analyzed (Participants) | 409
Number analyzed (hips) | 431
hips
  1 Year: Atrophy in any Cup Zones: No | 431
  1 Year: Atrophy in any Cup Zones: Yes | 0
  1 Year: Atrophy in any Cup Zones: N/A | 0
  1 Year: Atrophy in any Stem Zones: No | 428
  1 Year: Atrophy in any Stem Zones: Yes | 3
  1 Year: Atrophy in any Stem Zones: N/A | 0
  3 Years: Atrophy in any Cup Zones: number analyzed (Participants) | 392
  3 Years: Atrophy in any Cup Zones: number analyzed (hips) | 413
  3 Years: Atrophy in any Cup Zones: No | 413
  3 Years: Atrophy in any Cup Zones: Yes | 0
  3 Years: Atrophy in any Cup Zones: N/A | 0
  3 Years: Atrophy in any Stem Zones: number analyzed (Participants) | 392
  3 Years: Atrophy in any Stem Zones: number analyzed (hips) | 413
  3 Years: Atrophy in any Stem Zones: No | 411
  3 Years: Atrophy in any Stem Zones: Yes | 2
  3 Years: Atrophy in any Stem Zones: N/A | 0
  5 Years: Atrophy in any Cup Zones: number analyzed (Participants) | 338
  5 Years: Atrophy in any Cup Zones: number analyzed (hips) | 357
  5 Years: Atrophy in any Cup Zones: No | 357
  5 Years: Atrophy in any Cup Zones: Yes | 0
  5 Years: Atrophy in any Cup Zones: N/A | 0
  5 Years: Atrophy in any Stem Zones: number analyzed (Participants) | 338
  5 Years: Atrophy in any Stem Zones: number analyzed (hips) | 357
  5 Years: Atrophy in any Stem Zones: No | 357
  5 Years: Atrophy in any Stem Zones: Yes | 0
  5 Years: Atrophy in any Stem Zones: N/A | 0
  7 Years: Atrophy in any Cup Zones: number analyzed (Participants) | 315
  7 Years: Atrophy in any Cup Zones: number analyzed (hips) | 334
  7 Years: Atrophy in any Cup Zones: No | 334
  7 Years: Atrophy in any Cup Zones: Yes | 0
  7 Years: Atrophy in any Cup Zones: N/A | 0
  7 Years: Atrophy in any Stem Zones: number analyzed (Participants) | 315
  7 Years: Atrophy in any Stem Zones: number analyzed (hips) | 334
  7 Years: Atrophy in any Stem Zones: No | 332
  7 Years: Atrophy in any Stem Zones: Yes | 2
  7 Years: Atrophy in any Stem Zones: N/A | 0
  10 Years: Atrophy in any Cup Zones: number analyzed (Participants) | 278
  10 Years: Atrophy in any Cup Zones: number analyzed (hips) | 294
  10 Years: Atrophy in any Cup Zones: No | 293
  10 Years: Atrophy in any Cup Zones: Yes | 0
  10 Years: Atrophy in any Cup Zones: N/A | 1
  10 Years: Atrophy in any Stem Zones: number analyzed (Participants) | 278
  10 Years: Atrophy in any Stem Zones: number analyzed (hips) | 294
  10 Years: Atrophy in any Stem Zones: No | 290
  10 Years: Atrophy in any Stem Zones: Yes | 3
  10 Years: Atrophy in any Stem Zones: N/A | 1

6. Secondary Outcome: Radiographic Findings: Hypertrophy
Description: Number of participant hips with radiographic findings for hypertrophy indicated with a 'No', 'Yes', or 'N/A' (response not available) response at 1 year, 3 years, 5 years, 7 years, & 10 years for the following:
  * Hypertrophy in any Cup Zones
  * Hypertrophy in any Stem Zones
Time Frame: 1 years, 3 years, 5 years, 7 years, 10 years
Population: as for outcome 5
Measure: Count of Units; unit: hips
Units Other Than Participants: hips
Arm/Group | R3™ Acetabular System
Number analyzed (Participants) | 409
Number analyzed (hips) | 431
hips
  1 Year: Hypertrophy in any Cup Zones: No | 427
  1 Year: Hypertrophy in any Cup Zones: Yes | 4
  1 Year: Hypertrophy in any Cup Zones: N/A | 0
  1 Year: Hypertrophy in any Stem Zones: No | 399
  1 Year: Hypertrophy in any Stem Zones: Yes | 32
  1 Year: Hypertrophy in any Stem Zones: N/A | 0
  3 Years: Hypertrophy in any Cup Zones: number analyzed (Participants) | 392
  3 Years: Hypertrophy in any Cup Zones: number analyzed (hips) | 413
  3 Years: Hypertrophy in any Cup Zones: No | 412
  3 Years: Hypertrophy in any Cup Zones: Yes | 1
  3 Years: Hypertrophy in any Cup Zones: N/A | 0
  3 Years: Hypertrophy in any Stem Zones: number analyzed (Participants) | 392
  3 Years: Hypertrophy in any Stem Zones: number analyzed (hips) | 413
  3 Years: Hypertrophy in any Stem Zones: No | 350
  3 Years: Hypertrophy in any Stem Zones: Yes | 63
  3 Years: Hypertrophy in any Stem Zones: N/A | 0
  5 Years: Hypertrophy in any Cup Zones: number analyzed (Participants) | 338
  5 Years: Hypertrophy in any Cup Zones: number analyzed (hips) | 357
  5 Years: Hypertrophy in any Cup Zones: No | 357
  5 Years: Hypertrophy in any Cup Zones: Yes | 0
  5 Years: Hypertrophy in any Cup Zones: N/A | 0
  5 Years: Hypertrophy in any Stem Zones: number analyzed (Participants) | 338
  5 Years: Hypertrophy in any Stem Zones: number analyzed (hips) | 357
  5 Years: Hypertrophy in any Stem Zones: No | 347
  5 Years: Hypertrophy in any Stem Zones: Yes | 10
  5 Years: Hypertrophy in any Stem Zones: N/A | 0
  7 Years: Hypertrophy in any Cup Zones: number analyzed (Participants) | 315
  7 Years: Hypertrophy in any Cup Zones: number analyzed (hips) | 334
  7 Years: Hypertrophy in any Cup Zones: No | 334
  7 Years: Hypertrophy in any Cup Zones: Yes | 0
  7 Years: Hypertrophy in any Cup Zones: N/A | 0
  7 Years: Hypertrophy in any Stem Zones: number analyzed (Participants) | 315
  7 Years: Hypertrophy in any Stem Zones: number analyzed (hips) | 334
  7 Years: Hypertrophy in any Stem Zones: No | 325
  7 Years: Hypertrophy in any Stem Zones: Yes | 9
  7 Years: Hypertrophy in any Stem Zones: N/A | 0
  10 Years: Hypertrophy in any Cup Zones: number analyzed (Participants) | 278
  10 Years: Hypertrophy in any Cup Zones: number analyzed (hips) | 294
  10 Years: Hypertrophy in any Cup Zones: No | 293
  10 Years: Hypertrophy in any Cup Zones: Yes | 0
  10 Years: Hypertrophy in any Cup Zones: N/A | 1
  10 Years: Hypertrophy in any Stem Zones: number analyzed (Participants) | 278
  10 Years: Hypertrophy in any Stem Zones: number analyzed (hips) | 294
  10 Years: Hypertrophy in any Stem Zones: No | 281
  10 Years: Hypertrophy in any Stem Zones: Yes | 11
  10 Years: Hypertrophy in any Stem Zones: N/A | 2

7. Secondary Outcome: Radiographic Findings: Osteolysis
Description: Number of participant hips with radiographic findings for osteolysis greater than 2 millimeters in any cup or stem zones indicated with a 'No', 'Yes', or 'N/A' (response not available) response at 1 year, 3 years, 5 years, 7 years, & 10 years as the following:
  * Osteolysis > 2mm in any Cup Zones
  * Osteolysis > 2mm in any Stem Zones
Time Frame: 1 years, 3 years, 5 years, 7 years, 10 years
Population: as for outcome 5
Measure: Count of Units; unit: hips
Units Other Than Participants: hips
Arm/Group | R3™ Acetabular System
Number analyzed (Participants) | 409
Number analyzed (hips) | 431
hips
  1 Year: Osteolysis > 2mm in any Cup Zones: No | 403
  1 Year: Osteolysis > 2mm in any Cup Zones: Yes | 4
  1 Year: Osteolysis > 2mm in any Cup Zones: N/A | 24
  1 Year: Osteolysis > 2mm in any Stem Zones: No | 401
  1 Year: Osteolysis > 2mm in any Stem Zones: Yes | 5
  1 Year: Osteolysis > 2mm in any Stem Zones: N/A | 25
  3 Years: Osteolysis > 2mm in any Cup Zones: number analyzed (Participants) | 392
  3 Years: Osteolysis > 2mm in any Cup Zones: number analyzed (hips) | 413
  3 Years: Osteolysis > 2mm in any Cup Zones: No | 383
  3 Years: Osteolysis > 2mm in any Cup Zones: Yes | 6
  3 Years: Osteolysis > 2mm in any Cup Zones: N/A | 24
  3 Years: Osteolysis > 2mm in any Stem Zones: number analyzed (Participants) | 392
  3 Years: Osteolysis > 2mm in any Stem Zones: number analyzed (hips) | 413
  3 Years: Osteolysis > 2mm in any Stem Zones: No | 380
  3 Years: Osteolysis > 2mm in any Stem Zones: Yes | 7
  3 Years: Osteolysis > 2mm in any Stem Zones: N/A | 26
  5 Years: Osteolysis > 2mm in any Cup Zones: number analyzed (Participants) | 338
  5 Years: Osteolysis > 2mm in any Cup Zones: number analyzed (hips) | 357
  5 Years: Osteolysis > 2mm in any Cup Zones: No | 326
  5 Years: Osteolysis > 2mm in any Cup Zones: Yes | 6
  5 Years: Osteolysis > 2mm in any Cup Zones: N/A | 25
  5 Years: Osteolysis > 2mm in any Stem Zones: number analyzed (Participants) | 338
  5 Years: Osteolysis > 2mm in any Stem Zones: number analyzed (hips) | 357
  5 Years: Osteolysis > 2mm in any Stem Zones: No | 326
  5 Years: Osteolysis > 2mm in any Stem Zones: Yes | 4
  5 Years: Osteolysis > 2mm in any Stem Zones: N/A | 27
  7 Years: Osteolysis > 2mm in any Cup Zones: number analyzed (Participants) | 315
  7 Years: Osteolysis > 2mm in any Cup Zones: number analyzed (hips) | 334
  7 Years: Osteolysis > 2mm in any Cup Zones: No | 322
  7 Years: Osteolysis > 2mm in any Cup Zones: Yes | 2
  7 Years: Osteolysis > 2mm in any Cup Zones: N/A | 10
  7 Years: Osteolysis > 2mm in any Stem Zones: number analyzed (Participants) | 315
  7 Years: Osteolysis > 2mm in any Stem Zones: number analyzed (hips) | 334
  7 Years: Osteolysis > 2mm in any Stem Zones: No | 317
  7 Years: Osteolysis > 2mm in any Stem Zones: Yes | 7
  7 Years: Osteolysis > 2mm in any Stem Zones: N/A | 10
  10 Years: Osteolysis > 2mm in any Cup Zones: number analyzed (Participants) | 278
  10 Years: Osteolysis > 2mm in any Cup Zones: number analyzed (hips) | 294
  10 Years: Osteolysis > 2mm in any Cup Zones: No | 281
  10 Years: Osteolysis > 2mm in any Cup Zones: Yes | 1
  10 Years: Osteolysis > 2mm in any Cup Zones: N/A | 12
  10 Years: Osteolysis > 2mm in any Stem Zones: number analyzed (Participants) | 278
  10 Years: Osteolysis > 2mm in any Stem Zones: number analyzed (hips) | 294
  10 Years: Osteolysis > 2mm in any Stem Zones: No | 273
  10 Years: Osteolysis > 2mm in any Stem Zones: Yes | 9
  10 Years: Osteolysis > 2mm in any Stem Zones: N/A | 12

8. Secondary Outcome: Radiographic Findings: Radiolucent Lines (RLL)
Description: Number of participant hips with radiographic findings for radiolucent lines (RLL) greater than 2 millimeters in any cup or stem zones indicated with a 'No', 'Yes', or 'N/A' (response not available) response at 1 year, 3 years, 5 years, 7 years, & 10 years as the following:
  * RLL > 2mm in any Cup Zones
  * RLL > 2mm in any Stem Zones
Time Frame: 1 years, 3 years, 5 years, 7 years, 10 years
Population: as for outcome 5
Measure: Count of Units; unit: hips
Units Other Than Participants: hips
Arm/Group | R3™ Acetabular System
Number analyzed (Participants) | 409
Number analyzed (hips) | 431
hips
  1 Year: RLL > 2mm in any Cup Zones: No | 431
  1 Year: RLL > 2mm in any Cup Zones: Yes | 0
  1 Year: RLL > 2mm in any Cup Zones: N/A | 0
  1 Year: RLL > 2mm in any Stem Zones: No | 430
  1 Year: RLL > 2mm in any Stem Zones: Yes | 1
  1 Year: RLL > 2mm in any Stem Zones: N/A | 0
  3 Years: RLL > 2mm in any Cup Zones: number analyzed (Participants) | 392
  3 Years: RLL > 2mm in any Cup Zones: number analyzed (hips) | 413
  3 Years: RLL > 2mm in any Cup Zones: No | 413
  3 Years: RLL > 2mm in any Cup Zones: Yes | 0
  3 Years: RLL > 2mm in any Cup Zones: N/A | 0
  3 Years: RLL > 2mm in any Stem Zones: number analyzed (Participants) | 392
  3 Years: RLL > 2mm in any Stem Zones: number analyzed (hips) | 413
  3 Years: RLL > 2mm in any Stem Zones: No | 413
  3 Years: RLL > 2mm in any Stem Zones: Yes | 0
  3 Years: RLL > 2mm in any Stem Zones: N/A | 0
  5 Years: RLL > 2mm in any Cup Zones: number analyzed (Participants) | 338
  5 Years: RLL > 2mm in any Cup Zones: number analyzed (hips) | 357
  5 Years: RLL > 2mm in any Cup Zones: No | 356
  5 Years: RLL > 2mm in any Cup Zones: Yes | 1
  5 Years: RLL > 2mm in any Cup Zones: N/A | 0
  5 Years: RLL > 2mm in any Stem Zones: number analyzed (Participants) | 338
  5 Years: RLL > 2mm in any Stem Zones: number analyzed (hips) | 357
  5 Years: RLL > 2mm in any Stem Zones: No | 357
  5 Years: RLL > 2mm in any Stem Zones: Yes | 0
  5 Years: RLL > 2mm in any Stem Zones: N/A | 0
  7 Years: RLL > 2mm in any Cup Zones: number analyzed (Participants) | 315
  7 Years: RLL > 2mm in any Cup Zones: number analyzed (hips) | 334
  7 Years: RLL > 2mm in any Cup Zones: No | 333
  7 Years: RLL > 2mm in any Cup Zones: Yes | 1
  7 Years: RLL > 2mm in any Cup Zones: N/A | 0
  7 Years: RLL > 2mm in any Stem Zones: number analyzed (Participants) | 315
  7 Years: RLL > 2mm in any Stem Zones: number analyzed (hips) | 334
  7 Years: RLL > 2mm in any Stem Zones: No | 334
  7 Years: RLL > 2mm in any Stem Zones: Yes | 0
  7 Years: RLL > 2mm in any Stem Zones: N/A | 0
  10 Years: RLL > 2mm in any Cup Zones: number analyzed (Participants) | 278
  10 Years: RLL > 2mm in any Cup Zones: number analyzed (hips) | 294
  10 Years: RLL > 2mm in any Cup Zones: No | 292
  10 Years: RLL > 2mm in any Cup Zones: Yes | 1
  10 Years: RLL > 2mm in any Cup Zones: N/A | 1
  10 Years: RLL > 2mm in any Stem Zones: number analyzed (Participants) | 278
  10 Years: RLL > 2mm in any Stem Zones: number analyzed (hips) | 294
  10 Years: RLL > 2mm in any Stem Zones: No | 292
  10 Years: RLL > 2mm in any Stem Zones: Yes | 1
  10 Years: RLL > 2mm in any Stem Zones: N/A | 1

ADVERSE EVENTS:
Time Frame: Adverse Events were collected following implantation of the R3™ Acetabular System through 10 years.
Description: All adverse events (AE), regardless of their relationship to the study device were included in the safety analyses. Total participants at risk for each adverse event type (i.e., All Cause Mortality, Serious, and Other) indicates those with available AE data collected.
Arm/Group | R3™ Acetabular System
All-Cause Mortality (participants affected / at risk) | 37/478
Serious Adverse Events (participants affected / at risk) | 371/478
Other Adverse Events (participants affected / at risk) | 329/478
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R3™ Acetabular System (N=478)
Bursitis (Injury, poisoning and procedural complications) | 1 (1)
Cyst (Injury, poisoning and procedural complications) | 2 (2)
Death from unknown causes (Injury, poisoning and procedural complications) | 1 (1)
Deep Infection <6 weeks (Injury, poisoning and procedural complications) | 1 (1)
Deep Infection >6 weeks (Injury, poisoning and procedural complications) | 3 (4)
Deep Vein Thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Delayed Wound Healing (Injury, poisoning and procedural complications) | 4 (4)
Disturbance of skin sensation (Injury, poisoning and procedural complications) | 1 (1)
Elevated Metal Ions (Injury, poisoning and procedural complications) | 2 (3)
Fissure (Injury, poisoning and procedural complications) | 4 (4)
Groin pain, study hip side (Injury, poisoning and procedural complications) | 1 (1)
Hematoma, Hemarthrosis (Injury, poisoning and procedural complications) | 1 (1)
Inflammation (Injury, poisoning and procedural complications) | 2 (2)
Injury, poisoning, or consequence of external causes (Injury, poisoning and procedural complications) | 14 (14)
Leg Length Change (Injury, poisoning and procedural complications) | 7 (7)
Leg Pain (Injury, poisoning and procedural complications) | 1 (1)
Limp, study hip side (Injury, poisoning and procedural complications) | 1 (1)
Myalgia, muscle pain (Injury, poisoning and procedural complications) | 1 (1)
Operative side pain originating from other than study hip (Injury, poisoning and procedural complications) | 2 (2)
Pain in study hip (Injury, poisoning and procedural complications) | 10 (12)
Perioperative Fever (Injury, poisoning and procedural complications) | 2 (2)
Perioperative Pulmonary Embolism (Injury, poisoning and procedural complications) | 1 (1)
Post-op swelling of study leg (Injury, poisoning and procedural complications) | 2 (2)
Pseudotumor (Injury, poisoning and procedural complications) | 2 (2)
Reaction to metal debris/ metal allergy (Injury, poisoning and procedural complications) | 22 (22)
Tendonitis (Injury, poisoning and procedural complications) | 1 (1)
Trochanteritis (Injury, poisoning and procedural complications) | 2 (2)
Eye/Adnexa (Eye disorders) | 50 (65)
Death from unknown causes (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 43 (61)
Symptoms not otherwise defined (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Circulatory (Cardiac disorders) | 53 (83)
Death from unknown causes (Cardiac disorders) | 1 (1)
Nervous (Nervous system disorders) | 50 (61)
Pain, unknown etiology (Nervous system disorders) | 4 (4)
Symptoms not otherwise defined (Nervous system disorders) | 2 (2)
Death from unknown causes (General disorders) | 4 (4)
Pain, unknown etiology (General disorders) | 3 (4)
Lymphatic (Blood and lymphatic system disorders) | 3 (4)
Skin/Subcutaneous Tissue (Skin and subcutaneous tissue disorders) | 16 (17)
Ear/Mastoid Process (Ear and labyrinth disorders) | 4 (4)
Mental/behavioral (Psychiatric disorders) | 11 (12)
Digestive/Gastrointestinal (Hepatobiliary disorders) | 3 (3)
Bone Fracture- Femur (Musculoskeletal and connective tissue disorders) | 15 (16)
Digestive/Gastrointestinal (Musculoskeletal and connective tissue disorders) | 8 (8)
Dislocation (Musculoskeletal and connective tissue disorders) | 10 (14)
Heterotopic Ossification: Grade I (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular/Connective Tissue (Musculoskeletal and connective tissue disorders) | 28 (32)
Pain, unknown etiology (Musculoskeletal and connective tissue disorders) | 1 (1)
Skeletal (Musculoskeletal and connective tissue disorders) | 187 (298)
Superficial Infection Only (Musculoskeletal and connective tissue disorders) | 4 (4)
Symptoms not otherwise defined (Musculoskeletal and connective tissue disorders) | 1 (1)
Cancer, known origin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 57 (71)
Cancer, unknown type (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Death from unknown causes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Urinary (Renal and urinary disorders) | 38 (47)
Reproductive System (Reproductive system and breast disorders) | 17 (18)
Circulatory (Vascular disorders) | 46 (62)
Death from unknown causes (Vascular disorders) | 1 (1)
Hematologic/Immune System (Vascular disorders) | 12 (12)
Endocrine/Nutritional/Metabolic (Metabolism and nutrition disorders) | 21 (25)
Infection (Infections and infestations) | 21 (23)
Digestive/Gastrointestinal (Gastrointestinal disorders) | 51 (71)
Acetabular (Product Issues) | 1 (1)
Femoral (Product Issues) | 5 (5)
Femoral Component (Product Issues) | 6 (6)
Implant Failure (Product Issues) | 2 (2)
Other (Product Issues) | 1 (1)
Endocrine/Nutritional/Metabolic (Endocrine disorders) | 13 (13)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R3™ Acetabular System (N=478)
Back pain related to hip (Injury, poisoning and procedural complications) | 2 (2)
Bursitis (Injury, poisoning and procedural complications) | 6 (6)
Deep Infection <6 weeks (Injury, poisoning and procedural complications) | 1 (1)
Delayed Wound Healing (Injury, poisoning and procedural complications) | 1 (1)
Disturbance of skin sensation (Injury, poisoning and procedural complications) | 1 (1)
Ectopic Bone Formation (Injury, poisoning and procedural complications) | 1 (1)
Elevated Metal Ions (Injury, poisoning and procedural complications) | 23 (30)
Fissure (Injury, poisoning and procedural complications) | 2 (2)
Fluid Accumulation (Injury, poisoning and procedural complications) | 2 (2)
Groin pain, study hip side (Injury, poisoning and procedural complications) | 7 (7)
Hematoma, Hemarthrosis (Injury, poisoning and procedural complications) | 3 (3)
Hip Discomfort, soreness, or cramping, may be intermittent (Injury, poisoning and procedural complications) | 7 (7)
Hip Squeaking/Clicking/Popping/Snapping or other noise (Injury, poisoning and procedural complications) | 3 (3)
Inflammation (Injury, poisoning and procedural complications) | 1 (1)
Injury, poisoning, or consequence of external causes (Injury, poisoning and procedural complications) | 17 (20)
Leg Pain (Injury, poisoning and procedural complications) | 4 (4)
Limp, study hip side (Injury, poisoning and procedural complications) | 1 (1)
Myalgia, muscle pain (Injury, poisoning and procedural complications) | 1 (1)
Operative side pain originating from other than study hip (Injury, poisoning and procedural complications) | 1 (2)
Pain at Op site (Injury, poisoning and procedural complications) | 4 (4)
Pain in study hip (Injury, poisoning and procedural complications) | 25 (32)
Periaticular Calcification (Injury, poisoning and procedural complications) | 3 (3)
Perioperative Fever (Injury, poisoning and procedural complications) | 1 (1)
Post-op swelling of study leg (Injury, poisoning and procedural complications) | 4 (4)
Pseudotumor (Injury, poisoning and procedural complications) | 6 (6)
Psoas Tenopathy (Injury, poisoning and procedural complications) | 2 (2)
Reaction to metal debris/ metal allergy (Injury, poisoning and procedural complications) | 7 (7)
Stiffness (Injury, poisoning and procedural complications) | 2 (2)
Stress Shielding (Injury, poisoning and procedural complications) | 2 (2)
Tenderness in the trochanteric region (Injury, poisoning and procedural complications) | 2 (2)
Trendelenberg gait (Injury, poisoning and procedural complications) | 2 (2)
Trochanteritis (Injury, poisoning and procedural complications) | 10 (10)
Weakness in study leg (Injury, poisoning and procedural complications) | 2 (2)
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Eye/Adnexa (Eye disorders) | 13 (14)
Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 32 (36)
Symptoms not otherwise defined (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Circulatory (Cardiac disorders) | 16 (17)
Nervous (Nervous system disorders) | 37 (42)
Pain, unknown etiology (Nervous system disorders) | 8 (9)
Symptoms not otherwise defined (Nervous system disorders) | 1 (1)
Other (General disorders) | 2 (2)
Pain, unknown etiology (General disorders) | 6 (6)
Symptoms not otherwise defined (General disorders) | 1 (1)
Lymphatic (Blood and lymphatic system disorders) | 8 (8)
Other (Skin and subcutaneous tissue disorders) | 2 (2)
Skin/Subcutaneous Tissue (Skin and subcutaneous tissue disorders) | 36 (41)
Ear/Mastoid Process (Ear and labyrinth disorders) | 22 (26)
Special Sense (Ear and labyrinth disorders) | 2 (2)
Mental/behavioral (Psychiatric disorders) | 22 (23)
Bone Fracture- Femur (Musculoskeletal and connective tissue disorders) | 1 (1)
Cortical Thickening (Musculoskeletal and connective tissue disorders) | 1 (2)
Digestive/Gastrointestinal (Musculoskeletal and connective tissue disorders) | 3 (3)
Endocrine/Nutritional/Metabolic (Musculoskeletal and connective tissue disorders) | 6 (6)
Fracture-Subtrochanteric (Musculoskeletal and connective tissue disorders) | 1 (1)
Heterotopic Ossification- Generic Reporting (Musculoskeletal and connective tissue disorders) | 3 (3)
Heterotopic Ossification: Grade I (Musculoskeletal and connective tissue disorders) | 14 (14)
Muscular/Connective Tissue (Musculoskeletal and connective tissue disorders) | 47 (60)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, unknown etiology (Musculoskeletal and connective tissue disorders) | 8 (9)
Skeletal (Musculoskeletal and connective tissue disorders) | 175 (328)
Subluxation, no component specified (Musculoskeletal and connective tissue disorders) | 1 (1)
Superficial Infection Only (Musculoskeletal and connective tissue disorders) | 2 (2)
Symptoms not otherwise defined (Musculoskeletal and connective tissue disorders) | 2 (2)
Cancer, known origin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10)
Urinary (Renal and urinary disorders) | 27 (30)
Pain, unknown etiology (Reproductive system and breast disorders) | 1 (1)
Reproductive System (Reproductive system and breast disorders) | 11 (11)
Urinary (Reproductive system and breast disorders) | 1 (1)
Circulatory (Vascular disorders) | 27 (32)
Hematologic/Immune System (Vascular disorders) | 16 (17)
Symptoms not otherwise defined (Vascular disorders) | 1 (1)
Endocrine/Nutritional/Metabolic (Metabolism and nutrition disorders) | 18 (24)
Infection (Infections and infestations) | 13 (14)
Digestive/Gastrointestinal (Gastrointestinal disorders) | 40 (48)
Symptoms not otherwise defined (Gastrointestinal disorders) | 3 (3)
Femoral Component (Product Issues) | 2 (2)
Endocrine/Nutritional/Metabolic (Endocrine disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT04399928/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT04399928/SAP_001.pdf